CLINICAL TRIAL: NCT02818712
Title: Health-related Quality of Life and Comorbidities in Danish Patients With Idiopathic Pulmonary Fibrosis - a Nationwide Follow-up
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: IPF: HRQL, comorb and biomark
Record Dates: First submitted 2016-06-15; First posted 2016-06-30 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2020-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and EDTA-plasma is collected from all patients at 0, 6, 12, 24 and 36 months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with IPF

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a progressive lung disease with a high mortality. Health-related quality of life (HRQL) is impaired in patients with IPF. Little is known about the properties of recently developed HRQL questionnaires and about the longitudinal changes in HRQL, including factors with an impact on HRQL. Comorbidities have an impact on patients with IPF, but reports differ in incidence and prevalence. The impact of comorbidities on HRQL and disease progression has only been studied sparsely. Also, the association between biomarkers and disease progression need to be examined further.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of IPF
2. Signed informed consent

Exclusion Criteria:

1. Clinical, radiological or histological findings inconsistent with a diagnosis of IPF
2. Inability or unwillingness to adhere to the study
3. Active on lung transplantation list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident and prevalent patients with IPF in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Baseline, 6 months, 12 months, 24 months, 36 months
  Change in St. George's Respiratory Questionnaire
Health-related quality of life | Baseline, 2 weeks, 6 months, 12 months, 24 months, 36 months
  Change in St. George's Respiratory Questionnaire, IPF-specific
Health-related quality of life | Baseline, 2 weeks, 6 months, 12 months, 24 months, 36 months
  Changes in King's Brief Interstitial Lung Disease questionnaire
Number and type of comorbidities | Baseline
  Prevalence of comorbidities at baseline
Number and type of comorbidities | Change/incidence at 6 months, 12 months, 24 months and 36 months
  Incidence of new comorbidities after 6 months, 12 months, 24 months and 36 months

SECONDARY OUTCOMES:
Lung function tests | Baseline, 6 months, 12 months, 24 months, 36 months
  Change in forced vital capacity
Lung function tests | Baseline, 6 months, 12 months, 24 months, 36 months
  Change in diffusion capacity for carbon monoxide
6-minute walk test | Baseline, 6 months, 12 months, 24 months, 36 months
  Change in 6-minute walk test
Progression in serum/plasma biomarker levels | Baseline, 6 months, 12 months, 24 months, 36 months
  Increase or decrease in serum/plasma biomarker levels
Health-related quality of life | Baseline, 6 months, 12 months, 24 months, 36 months
  Change in Short Form 36
Health-related quality of life | Baseline, 6 months, 12 months, 24 months, 36 months
  Changes in University of California San Diego Shortness Of Breath Questionnaire
Disease progression | Baseline, 12 months, 24 months, 36 months
  Change in interstitial changes on high resolution CT-scan (HRCT)
Disease progression | Baseline, 6 months, 12 months, 24 months, 36 months
  Changes in number of acute exacerbations
Disease progression | Baseline, 6 months, 12 months, 24 months, 36 months
  Changes in use of supplementary oxygen

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aarhus University Hosptial, Aarhus C
  - Gentofte Hospital, Hellerup
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hansen AH, Breisnes HW, Prior TS, Hilberg O, Rasmussen DGK, Genovese F, Lukassen MV, Svensson B, Langholm LL, Manon-Jensen T, Karsdal MA, Leeming DJ, Bendstrup E, Sand JMB. A serologically assessed neo-epitope biomarker of cellular fibronectin degradation is related to pulmonary fibrosis. Clin Biochem. 2023 Aug;118:110599. doi: 10.1016/j.clinbiochem.2023.110599. Epub 2023 Jun 19. PMID 37343745
- [Derived] Prior TS, Hoyer N, Hilberg O, Shaker SB, Davidsen JR, Bendstrup E. Responsiveness and minimal clinically important difference of SGRQ-I and K-BILD in idiopathic pulmonary fibrosis. Respir Res. 2020 Apr 21;21(1):91. doi: 10.1186/s12931-020-01359-3. PMID 32316976
- [Derived] Prior TS, Hilberg O, Shaker SB, Davidsen JR, Hoyer N, Birring SS, Bendstrup E. Validation of the King's Brief Interstitial Lung Disease questionnaire in Idiopathic Pulmonary Fibrosis. BMC Pulm Med. 2019 Dec 19;19(1):255. doi: 10.1186/s12890-019-1018-0. PMID 31856786
- [Derived] Prior TS, Hoyer N, Shaker SB, Davidsen JR, Yorke J, Hilberg O, Bendstrup E. Validation of the IPF-specific version of St. George's Respiratory Questionnaire. Respir Res. 2019 Aug 28;20(1):199. doi: 10.1186/s12931-019-1169-9. PMID 31462235